CLINICAL TRIAL: NCT00633308
Title: Phosphorus and Calcium Removal During Long Hemodialysis Treatment Sessions
Acronym: hemodialysis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No coordinator available to work on study.
Sponsor: Indiana University (Other)
Responsible Party: Michael Kraus, M.D., Indiana University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NxStage LongHD
Record Dates: First submitted 2008-02-21; First posted 2008-03-12 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Kidney Failure
Keywords: hemodialysis
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Long hemodialysis
  Interventions: Device: NxStage System One (NxStage Medical, Lawrence, MA)

INTERVENTIONS:
Device: NxStage System One (NxStage Medical, Lawrence, MA) — Each patient will be studied on 4 separate occasions. The study sessions are longer than routine daily hemodialysis therapy using the System One.
  Other Names: The System One (NxStage Medical, Lawrence, MA)

SUMMARY:
The purpose of this sudy is to determined the effect of dialysate volume and treatment time on phosphate and calcium removal in stage V chronickidney disease patients treated by hemodialysis using the System One (NxStage Medical, Lawrence, MA)

DETAILED DESCRIPTION:
Ten patients will be recruited from those routinely treated in-center or at home using the Systerm One at the clinical centers. Each patient will be studiesd on 4 separate occastions. Treatments under the following conditions will each be performed on each study patient, at least one week apart:

1. Treatment for 8 hrs uding 40L of dialysate
2. Treatment for 8 hrs using 60L of dialysate
3. Treatment for 5 hrs using 40L of dialysate
4. Treatment for 5 hrs using 60L of dialysate

Blood samples will be collected and assayed for the concentrations of urea, phosphate, calcium, bicarbonate, beta-2-microglobulin and albumin using standard assays.

ELIGIBILITY:
Inclusion Criteria:

* Stage V chronic kidney patients with minimal or no residual renal functin

Exclusion Criteria:

* Medically unstable
* Hematocrit less than 28%
* Hepatitis B positive, hepatitis C positive or HIV positive
* Pregnant women
* Minors below 18 years of age
* Active psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2010-01 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
the effect of dialysate volume and treatment time on phosphage and calcium removal | 4 treatments

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kraus, M.D., Principal Investigator — Indiana University